CLINICAL TRIAL: NCT01334437
Title: Blood Test for Ovarian Cancer Associated Auto Antibodies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eventus Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EventusDx_ovary_2011ver2
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Ovarian Cancer
Keywords: blood test; ovarian cancer; Associated Auto Antibodies
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Intend of use: A blood test for Cancer Associated Antibodies (CAAA) is an aid in initial diagnosis of ovarian cancer in women with suspected ovarian pathology as detected by primary diagnostic techniques.

Test Description: Blood is collected from patients and serum/plasma is tested for the presence of CAAA on experimental test kit.

Objectives: To assess the effectiveness of the CAAA test.

Target Population:

The study population will include women that have been diagnosed with suspected ovarian cancer (OC), verified by pathology/cytology as patients, women with suspected ovarian cancer but verified by pathology/cytology as non-cancers and a control set of blood samples will be collected from age matched women with no history of cancer.

Structure: Women that will be enrolled for the study will be checked for the presence of CAAAb, and the results of the CAAAb test will be compared to the pathology submitted by the physicians in the participating centers for the patient population and to the clinical history for the control population.

Sample Size: The investigators will collect at least 50 patients verified by pathology/cytology and for each patient at least two aged matched healthy controls and two aged matched suspected but verified as non-cancers. Total amount at least 250 samples.

(Multi center study, statistical rationale provided below).

Primary Effectiveness Variables: The effectiveness of the test will be defined by the specificity of the test conditionally that the sensitivity is not lower than a pre-defined level of 95%.

Endpoint: The endpoint of this study is to show that the effectiveness is higher than 50%.

Clinical Monitor: For each site a dedicated CRO will be appointed to monitor the clinical trials. All data will be stored in a protected internet-based database, and any changes of the data will be traced and recorded.

DETAILED DESCRIPTION:
Since the mutations of a normal cell that lead to a malignancy, involves changes in the structure and function of the cells, it could be assumed that the immune system has recognized some of these changes as antigenic determinates that should be responded against. For many years, investigators tried to distinguish between cancer patients and healthy population by the difference in specific autoantibodies level. In the healthy population, a baseline of the amount of autoantibodies was determined, and the patient population had to have a statistically significant higher level of autoantibodies. The presence of autoantibodies in all population in different levels made it very difficult to find these specifically discriminating antibodies. To date, no specific autoantibody is distinguishing solely between healthy and cancer patients (as opposed to autoimmune diseases, where specific autoantibodies can be found in very high levels in patients only).

Our work assumes that specific Autoantibodies expression level should be altered in cancer, and thus these changes can indicate the presence / absence of cancer.

In this experiment protocol, we are checking for changes in expression levels of specific autoantibodies of women with ovarian pathology compared to women without cancer.

The CAAA test is comprised of a blood collection and processing step followed by detection of specific auto antibodies with an ELISA based assay and a mathematical processing, with a subsequent classification of the results as "positive" or "negative" for ovarian cancer.

The study population includes those women that are scheduled for a pathological or cytological confirmation either by a surgical procedure (laparoscopy/laparotomy) or any kind of biopsy or cytology, prior to any anti-cancer treatment and aged matched controls. The clinical suspicion includes one of the following: Pelvic mass/cyst (by pelvic examination and/or imaging techniques), and/or high CA-125 levels, and/or ascites, and/or due to incidental finding of distant metastasis. Final verification ("true positive" or "true negative") will be done in relation to pathology/cytology results only or for healthy women in relation to clinical history.

Subject Selection Suspected ovarian cancer women(patients and non-cancers women) - Inclusion criteria - all of the following

* 18 years or over.
* Patients suspected of ovarian pathology. The clinical suspicion will include one of the following: Pelvic mass/cyst (by pelvic examination and/or other imaging techniques), and/or high CA-125 levels, and/or ascites, and/or due to incidental finding of distant metastasis. Final analysis will be done in relation to pathology/cytology results only.
* Patients scheduled laparotomy/laparoscopy/surgery, ideally before any of the above.

Suspected ovarian cancer women(patients and non-cancers women) - Exclusion criteria: any of the following

* Less than 18 years of age
* Hematological malignancies
* Autoimmune disorders diagnosed patients.
* Previous or current tumors
* Patients under active chemotherapy treatment

Suspected ovarian cancer patients - final classification

• The "true positive" group consists of all sequential patients that satisfy inclusion criteria and are positive for ovarian cancer by pathology results. The "true negative" group consists of sequential patients that satisfy inclusion criteria and are negative for ovarian cancer by pathology results.

This study will be based on multi-centers participation. The minimum number of sites for the study is 2.

The current study is a single blind prospective validation study, involving all consecutive suspected ovarian pathology women being scheduled for biopsy/surgery during the study duration, having pathology/cytology ovarian cancer (true positive) and XXX number of women having negative ovarian pathology/cytology results (true negative)and healthy women. The purpose of the study is to evaluate the effectiveness of the CAAA test.

The effectiveness of the study is defined as the specificity of the CAAA test for a pre defined sensitivity of 95%.

The study will evaluate the sensitivity of CAAA test to show that it is not below the declared level of 95%.

According to current medical publications, we assume that the study population will include about 10-20% of true positive cancer cases.

As of today, large proportion of the suspected patients was only diagnosed by final pathology of the laparoscopy/surgery. In this study, the true positive and true negative cases (as verified by pathology) will be compared to the CAAA test results.

Study Procedure Subjects clinical information acquired from the patient's medical file, including age, medical history and results of tests done leading to the diagnostic evaluation of ovarian cancer will be recorded on the appropriate, bar-coded, pre-study case report forms .The reports will be electronic via a dedicated and secured internet site, any changes in the database will be recorded and will be traceable. The study is anonymous and the Department will keep the name of the patient without reveling it to investigators and to the study sponsor.

The doctor/ nurse/ phlebotomist will collect a heparin vacuum/serological tube (about 8ml), label (bar-code) them. The blood handling laboratory will collect serum/plasma and the serum will be kept frozen at -80C.

ELISA based tests for the detection of Auto Antibodies relative expression ratios, will be conducted on each sample according to the lab protocol . The samples will be tested for response to the antigens that have been identified on a previous training set. All the data will be permanently recorded directly into a dedicated computer. For each sample all antibody results will be put into the coded patient file. A mathematical algorithm will determine if the sample is positive or negative.

The final pathology will be compared with the CAAA test results. The results will be analyzed by a statistician with expertise in cancer population studies.

The current study is a blind prospective validation study, involving all consecutive suspected ovarian pathology subjects being scheduled for biopsy/surgery/cytology during the study duration. The purpose of the study is to assess the sensitivity and specificity of the CAAA test for detection ovarian cancer in women scheduled for biopsy/surgery/cytology.

Subjects will be screened for potential participation in the study, according to the inclusion and exclusion criteria.

The data will include parameters of the clinical and pathological/cytological state of the subjects and results of CAAA ELISA.

There are two goals of the study. To test that the sensitivity of CAAA is not below the pre-defined level. To evaluate the specificity of CAAA test. Statistical Hypothesis The main condition determining the sample size is to validate that the sensitivity of the test is not lower than the predefined level. The classification rule was established in such a way that the sensitivity in the teaching sample was 100%. We assume that the real sensitivity is not lower that 99%.

Null Hypothesis: The sensitivity of the test is not higher than 95%. A database management system shall be designed and maintained, including screen preparation, and edit check programming. Pre-entry and post-entry quality control of the clinical data shall be performed at each data entry center. All ELISA test results will be uploaded to the database via an internet based interface, and will be locked against further changes. In order to change ELISA test results, unlocking of the database requires consent from the local CRO, the sponsor and the site physician. Unlocking will be done only by the webmaster, and will be recorder in the tracing system component, and in a hard copy held both by the sponsor and the CRO in the site.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over.
* Patients suspected of ovarian pathology. The clinical suspicion will include one of the following: Pelvic mass/cyst (by pelvic examination and/or other imaging techniques), and/or high CA-125 levels, and/or ascites, and/or due to incidental finding of distant metastasis. Final analysis will be done in relation to pathology/cytology results only.
* Patients scheduled laparotomy/laparoscopy/surgery, ideally before any of the above.

Exclusion Criteria:

* Less than 18 years of age
* Hematological malignancies
* Autoimmune disorders diagnosed patients.
* Previous or current tumors
* Patients under active chemotherapy treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include women that have been diagnosed with suspected ovarian cancer (OC), verified by pathology/cytology as patients, women with suspected ovarian cancer but verified by pathology/cytology as non-cancers and a control set of blood samples will be collected from age matched women with no history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants in each of the clinicaly defined groups (OC, suspected and control). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Lavie, Professor, Principal Investigator — Carmel Hospital
Locations (1):
- "Carmel" Medical Center, Haifa, Israel